CLINICAL TRIAL: NCT02880124
Title: Ingestion of Maple Products During Exercise: Effects on Energy Metabolism and Time-trial Performance
Brief Title: Maple Products and Exercise Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: Fédération des producteurs acéricoles du Québec (Unknown)
Responsible Party: Principal Investigator, Jonathan Tremblay, Professeur agrégé, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16-088-CERES-P
Record Dates: First submitted 2016-07-30; First posted 2016-08-26 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Carbohydrate Ingestion; Fuel Selection; Athletic Performance
Keywords: Isotope Labeling, Stable; Exercise, Physical; Calorimetry, Indirect; Athletic Performance; Sugar Maple
MeSH Terms: conditions — Motor Activity | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Maple syrup (Experimental): A maple syrup solution of 6% carbohydrate per volume labeled with 13C-sucrose will be ingested 30 min prior to starting exercise and every 30 min thereafter (solution ingestion), until 2h of the constant load cycling exercise is completed. Starting 4 min before each solution ingested over the protocol, indirect respiratory calorimetry, expired gas sampling, blood sampling will occur. After completing the 2h of exercise, subjects will be given a few minutes of rest (5-min) during which the catheter will be removed, after which the 20-km time trial will be initiated on the same ergometer. Palatability of the solution will be assessed after the first ingestion and after ingesting the last solution. Gastrointestinal symptoms will be assessed after the time trial.
  Interventions: Dietary Supplement: Solution ingestion; Behavioral: Constant load cycling; Procedure: Expired gas sampling; Procedure: Indirect respiratory calorimetry; Other: Palatability; Other: Gastrointestinal; Procedure: Blood sampling; Behavioral: Time trial
- Maple sap (Experimental): A maple sap solution of 6% carbohydrate per volume labeled with 13C-sucrose will be ingested 30 min prior to starting exercise and every 30 min thereafter (solution ingestion), until 2h of the constant load cycling exercise is completed. Starting 4 min before each solution ingested over the protocol, indirect respiratory calorimetry, expired gas sampling, blood sampling will occur. After completing the 2h of exercise, subjects will be given a few minutes of rest (5-min) during which the catheter will be removed, after which the 20-km time trial will be initiated on the same ergometer. Palatability of the solution will be assessed after the first ingestion and after ingesting the last solution. Gastrointestinal symptoms will be assessed after the time trial.
  Interventions: Dietary Supplement: Solution ingestion; Behavioral: Constant load cycling; Procedure: Expired gas sampling; Procedure: Indirect respiratory calorimetry; Other: Palatability; Other: Gastrointestinal; Procedure: Blood sampling; Behavioral: Time trial
- Glucose (Active Comparator): A glucose solution of 6% carbohydrate per volume labeled with 13C-sucrose will be ingested 30 min prior to starting exercise and every 30 min thereafter (solution ingestion), until 2h of the constant load cycling exercise is completed. Starting 4 min before each solution ingested over the protocol, indirect respiratory calorimetry, expired gas sampling, blood sampling will occur. After completing the 2h of exercise, subjects will be given a few minutes of rest (5-min) during which the catheter will be removed, after which the 20-km time trial will be initiated on the same ergometer. Palatability of the solution will be assessed after the first ingestion and after ingesting the last solution. Gastrointestinal symptoms will be assessed after the time trial.
  Interventions: Dietary Supplement: Solution ingestion; Behavioral: Constant load cycling; Procedure: Expired gas sampling; Procedure: Indirect respiratory calorimetry; Other: Palatability; Other: Gastrointestinal; Procedure: Blood sampling; Behavioral: Time trial
- Sport drink (Active Comparator): A Gatorade (TM) solution of 6% carbohydrate per volume labeled with 13C-sucrose will be ingested 30 min prior to starting exercise and every 30 min thereafter (solution ingestion), until 2h of the constant load cycling exercise is completed. Starting 4 min before each solution ingested over the protocol, indirect respiratory calorimetry, expired gas sampling, blood sampling will occur. After completing the 2h of exercise, subjects will be given a few minutes of rest (5-min) during which the catheter will be removed, after which the 20-km time trial will be initiated on the same ergometer. Palatability of the solution will be assessed after the first ingestion and after ingesting the last solution. Gastrointestinal symptoms will be assessed after the time trial.
  Interventions: Dietary Supplement: Solution ingestion; Behavioral: Constant load cycling; Procedure: Expired gas sampling; Procedure: Indirect respiratory calorimetry; Other: Palatability; Other: Gastrointestinal; Procedure: Blood sampling; Behavioral: Time trial
- Trace (Placebo Comparator): A solution containing stevia (sugar substitute) and trace amounts of glucose (3g) labeled with 13C-sucrose will be ingested 30 min prior to starting exercise and every 30 min thereafter (solution ingestion), until 2h of the constant load cycling exercise is completed. Starting 4 min before each solution ingested over the protocol, indirect respiratory calorimetry, expired gas sampling, blood sampling will occur. After completing the 2h of exercise, subjects will be given a few minutes of rest (5-min) during which the catheter will be removed, after which the 20-km time trial will be initiated on the same ergometer. Palatability of the solution will be assessed after the first ingestion and after ingesting the last solution. Gastrointestinal symptoms will be assessed after the time trial.
  Interventions: Dietary Supplement: Solution ingestion; Behavioral: Constant load cycling; Procedure: Expired gas sampling; Procedure: Indirect respiratory calorimetry; Other: Palatability; Other: Gastrointestinal; Procedure: Blood sampling; Behavioral: Time trial

INTERVENTIONS:
Dietary Supplement: Solution ingestion — Subjects will be required to ingest 2 litres of the experimental solution, spread over the 2 hours of exercise. A first ingestion of 572 mL of solution will be made at rest, 30 minutes before starting exercise, and 286 mL will be ingested immediately before the start of exercise and every 30 minutes during the exercise period.
Behavioral: Constant load cycling — Subjects will be required to perform 2 hours of cycling exercise at a power output eliciting 60% of VO2max.
Procedure: Expired gas sampling — Subjects will be asked, twice, to provide a forced expiration into a 10 mL plastic tube in order to collect a sample expired gases. This procedure will be done immediately before blood sampling and ingestion of the solution, every 30 minutes.
Procedure: Indirect respiratory calorimetry — A mouthpiece and nose plug will be placed on the subject and expired gases will be analyzed by a metabolic cart during 3 minutes. This procedure will be done immediately before expired gas collection, blood sampling and ingestion of the solution, every 30 minutes.
Other: Palatability — Subjects will be asked to fill out a short form on the palatability of the solution ingestion, after ingesting the first solution and at the end of exercise, after ingestion the last solution.
Other: Gastrointestinal — At the end of the time trial, subjects will be asked to fill out a short form on gastrointestinal issues they might have had during experimentation.
Procedure: Blood sampling — A catheter will be inserted in an antecubital vein and a saline solution will be continuously perfused to maintain the vessel open. 15 mL of blood will be collected every 30 minutes, immediately before ingesting the solution.
Behavioral: Time trial — Subjects will be required to complete a simulated 20-km time trial on the cycle ergometer set in linear mode (where resistance is proportional to pedalling cadence), starting at 70% of the peak power output for the cadence spontaneously adopted by the subject during 2 hours of exercise.

SUMMARY:
The purpose of this study is to compare the acute metabolic responses and time-trial performance following the ingestion of carbohydrate solutions containing either maple syrup, maple sap, corn syrup, a commercial sport drink or water.

DETAILED DESCRIPTION:
The study will require 4 meetings for each subject: a 30-minute meeting to explain the project; a meeting of 2 hours (glucose tolerance test, at rest); a one-hour meeting (maximum oxygen consumption test (VO2max) during an exercise conducted on an electromagnetically braked cycle ergometer, and a meeting of about 4 hours for experimentation (120-min exercise on a stationary bicycle with ingestion of a solution carbohydrates or sweetened water, and a 20-km time trial).

Visit #1 - Pre-participation (screening visit) Following an initial contact by phone or email, the subject will be invited to individual meetings which will last about 15 minutes. During the meeting, one of the project managers will check the eligibility of the potential subject in the study and, if eligible, will present him the details of the protocol specifying the discomforts and risks involved. The participant will be required to fill a Physical Activity Readiness Questionnaire (PAR-Q) and will be given a copy of the consent form. We will request the name and contact details of a person to contact in case of emergency, this information will be recorded and preserved in the subject matter. A period of at least three days will be allocated to make the decision whether to participate in the study or not. If the participant decides to participate in the study, he will be invited for the second visit (oral glucose tolerance test) and on this occasion will sign the consent form.

Visit #2 - Oral glucose tolerance test (OGTT) This test will be performed at Exercise Physiology Laboratory at the Department of kinesiology from the University of Montreal under the procedure commonly used for these tests. This procedure requires the ingestion of 300 mL of water containing 75 g of glucose in the morning (around 8am) after 12 hours of fasting, and blood samples and on the tip of a finger at 0, 60 and 120 minutes for the measurement of blood glucose. Subjects with higher blood glucose than 5 mmol/L before ingestion of glucose and greater than 8 mmol/L after ingestion (60 or 120 min) will not be considered for the study. These glucose tolerance standards are more stringent than those of the World Health Organization, because the objective of this test is not a diagnosis on glucose tolerance or a prognosis of its future development, but just n include in the study subjects who have good glucose tolerance.

Visit #3 - Maximum oxygen uptake testing: cycling VO2max This test will be conducted in the Exercise Physiology Laboratory at the Department of kinesiology from the University of Montreal. Exercise involves pedaling a stationary bike at a power output (resistance) gradually increasing until reaching VO2max. During the execution of the test, the subject is wearing surface electrodes to measure heart rate, a mouthpiece and nose clip to measure the volume of expired gas as well as the oxygen and carbon dioxide content to determine the consumption oxygen and carbon dioxide production. This type of testing is routinely used in our laboratory. The test can be stopped at any time by the will of the subject. For this test, guidelines established by the Exercise Physiology Laboratory at the Department of kinesiology from the University of Montreal will be followed. These guidelines are based on recommendations of ethics and safety of the "American College of Sports Medicine".

4- Experimentation The tests will be conducted at the Exercise Physiology Laboratory at the Department of kinesiology from the University of Montreal. The exercise is carried out on stationary cycle ergometer. It lasts 120 minutes at a power output corresponding to 60% of the VO2max obtained during the maximal test. A volume of a carbohydrate solution (120 g, 6% carbohydrate by volume) or sweetened water will be administered to the subject before (571 mL) and during exercise (286 mL every 30 minutes). The following solutions will be administered in a balanced, randomized, double-blind model: maple sap, maple syrup, glucose, a commercial sports drink and water with a glucose trace (0.001% carbohydrate by volume). Under conditions where only a trace of water or glucose are administered, a natural sweetener (stevia) will be added to obtain a sweet taste similar to other conditions. Carbohydrate solutions will all be artificially enriched in 13C. The volume ingested after 30 minutes of exercise will be artificially enriched in deuterium (D2O, 8g incorporated in the ingestion of 286 mL).

ELIGIBILITY:
Inclusion Criteria:

* Low alcohol consumption (<3 drinks/week)
* Not regularly taking medication for a known pathology
* Regularly practices endurance sports (cycling, running, etc.)

Exclusion Criteria:

* Intolerant to glucose (according to WHO standards)
* Musculoskeletal injury or illness affecting exercise performance
* Failure to respect protocol guidelines (diet, exercise prior to experimentation, etc.)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Exogenous carbohydrate oxidation | Every 30 minutes during the exercise protocol, during 3 minutes of expired gas collection.
  Measured by indirect respiratory calorimetry combined with tracer techniques.
Exercise performance in the 20-km time trial | At the end of 2 hours of exercise
  Duration to complete distance and mean power sustained during the performance

SECONDARY OUTCOMES:
Blood insulin concentration | Every 30 minutes during the exercise protocol
  Blood is sampled using a venous catheter over about 60 seconds. Following centrifugation to extract the plasma, a small sample is used to measure insulin concentration.
Blood glucose concentration | Every 30 minutes during the exercise protocol
  Blood is sampled using a venous catheter over about 60 seconds. Following centrifugation to extract the plasma, a small sample is used to measure glucose concentration.
Blood free fatty acid concentration | Every 30 minutes during the exercise protocol
  Blood is sampled using a venous catheter over about 60 seconds. Following centrifugation to extract the plasma, a small sample is used to measure free fatty acid concentration.
Blood lactate concentration | Every 30 minutes during the exercise protocol
  Blood is sampled using a venous catheter over about 60 seconds. Following centrifugation to extract the plasma, a small sample is used to measure lactate concentration.
Muscle glycogen oxidation | Every 30 minutes during the exercise protocol, during 3 minutes of expired gas collection.
  Measured by indirect respiratory calorimetry combined with tracer techniques.
Oxidation of glucose released by the liver | Every 30 minutes during the exercise protocol, during 3 minutes of expired gas collection.
  Measured by indirect respiratory calorimetry combined with tracer techniques. Average of 3 minutes of steady-state expired gas collection.
Total carbohydrate oxidation | Every 30 minutes during the exercise protocol, during 3 minutes of expired gas collection.
  Measured by indirect respiratory calorimetry.

OTHER OUTCOMES:
Palatability score | Within 5 minutes after the first ingestion and within 5 minutes after the last ingestion.
  Score computed from ratings on a visual analog scale.
Score of gastrointestinal symptoms | Within 5 minutes after the end of exercise
  Score computed from ratings on a visual analog scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Tremblay, Ph.D., Principal Investigator — Université de Montréal
Locations (1):
- Centre d'éducation physique et sportive de l'Université de Montréal (CEPSUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lavoie L, Tremblay J. Ingestion of maple-based and other carbohydrate sports drinks: effect on sensory perceptions during prolonged exercise. J Int Soc Sports Nutr. 2020 Dec 9;17(1):63. doi: 10.1186/s12970-020-00384-3. PMID 33298104